CLINICAL TRIAL: NCT00121732
Title: A Phase 1, Two-Arm, Open-Label Study of E7974 Administered on Days 1, 8, and 15 of a 28-Day Cycle and Days 1 and 8 of a 21-Day Cycle in Patients With Solid Malignancies
Brief Title: An Open-Label Study of E7974 Administered on Days 1, 8, and 15 of a 28-Day Cycle and Days 1 and 8 of a 21-Day Cycle in Patients With Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7974-A001-101
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumor Malignancies, Cancer
MeSH Terms: conditions — Neoplasms | interventions — E 7974

ARMS (2):
- A (Experimental)
  Interventions: Drug: E7974
- B (Experimental)
  Interventions: Drug: E7974

INTERVENTIONS:
Drug: E7974 — Maximum tolerated dose = 0.15 mg/m^2 administered on Days 1, 8, 15 of 28-day cycle.
  Arms: A
Drug: E7974 — Maximum tolerated dose = 0.37 mg/m^2 administered on Days 1 and 8 of 21-day cycle.
  Arms: B

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of E7974 administered as an intravenous bolus dose on Days 1, 8, and 15 of a 28-day cycle (Arm A) or on Days 1 and 8 of a 21-day cycle (Arm B) to patients with solid tumors that have progressed following effective therapy or for which no effective therapy exists.

DETAILED DESCRIPTION:
This is a two-arm, open-label, non-randomized, dose-escalation study to determine the MTD of E7974 administered as an intravenous bolus dose on Days 1, 8, and 15 of a 28-day cycle (Arm A) or on Days 1 and 8 of a 21-day cycle (Arm B) to patients with solid tumors that have progressed following effective therapy or for which no effective therapy exists. Response and progression will be evaluated in this study using Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the inclusion criteria and none of the exclusion criteria will be eligible for entry into the study:

1. Patients must have a pathologically diagnosed, histologically or cytologically confirmed solid tumor that has progressed following effective therapy or for which no effective therapy exists (including surgery or radiation therapy).
2. Patients must be >= 18 years of age.
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.
4. Patients must have a life expectancy of >= 3 months.
5. Patients must have adequate renal function as evidenced by serum creatinine <= 1.5 mg/dL or creatinine clearance >= 40 mL/minute (min).
6. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count >= 1,500/µL, hemoglobin of >= 9 g/dL (may be transfused), and platelet count (not transfused) >= 100,000/µL.
7. Patients must have adequate liver function as evidenced by bilirubin <= 1.5 mg/dL and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3 times the upper limits of normal (ULN), unless related to liver involvement by tumor, in which case <= 5.0 times ULN.
8. Patients must be willing and able to sign written informed consent and be able to comply with the study protocol for the duration of the study.
9. Patients must be willing and able to undergo blood draw and urine sampling for PK in Cycle 1.
10. Patients may have either measurable or non-measurable disease.

Exclusion Criteria:

The presence of one or more of the following criteria will disqualify a patient from enrollment in the study:

1. Patients who have received chemotherapy within three weeks of E7974 treatment start (6 weeks for a nitrosourea).
2. Patients who have not recovered from any chemotherapy-related or other therapy-related toxicity to <= Grade 1 at study entry (excluding Grade 2 alopecia).
3. Patients who have received radiotherapy <= 3 weeks prior to study enrollment, whose marrow exposure has exceeded 25% and who have not recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia).
4. Patients who have had major surgery without full recovery or major surgery within three weeks of E7974 treatment start.
5. Patients with primary brain tumors or metastasis at study entry must have controlled them for >= 1 month by previous treatment, including radiation therapy and corticosteroids.
6. Women who are pregnant or breastfeeding.
7. Women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test.
8. Women of childbearing potential unless (1) surgically sterile, (2) physiologically postmenopausal for > 12 months, or (3) using adequate measures (including barrier methods) of contraception.
9. Fertile men or their partners who are not willing to use contraception.
10. Patients who have a positive history for Human Immunodeficiency Virus (HIV) and/or have active hepatitis B or active hepatitis C at study entry.
11. Patients with severe, uncontrolled intercurrent illness or infection.
12. Patients with medically uncontrolled cardiovascular illness defined as unstable angina, >= symptomatic Grade II New York Heart Association (NYHA) Classification congestive heart failure (CHF), or myocardial infarction within six months prior to study entry.
13. Patients who have received organ allografts requiring immunosuppressive therapy.
14. Patients who have received investigational drugs including immunotherapy, gene therapy, hormone therapy, biologic therapy, or chemotherapy within the three-week period prior to E7974 treatment start; patients must have recovered from any previous major therapy-related toxicities (Grade 3 or 4) to <= Grade 1 at study entry.
15. Patients with a current history of peripheral neuropathy > CTC Grade 2 (e.g., diabetic or chemotherapy-induced neuropathy).
16. Patients with a history of uncontrolled seizures.
17. Patients with marked baseline prolongation of QT/QTc interval (QTc interval >470) using the Fridericia method as the main method of QTc analysis.
18. Patients with other significant diseases or disorders that, in the Investigator's opinion, would exclude them from the study.
19. Patients with allergy or hypersensitivity to hemiasterlin based product or analogue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of E7974 in patients with solid malignancies. | Duration of each cycle will be 28 or 21 days; patients will attend a follow-up visit 30 days after last study treatment. Follow-up for safety and efficacy will occur 6 months after the last patient is accrued to the study.

SECONDARY OUTCOMES:
1) Assess E7974 for safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD); 2) Evaluate the correlation of AUC with clinical toxicity and efficacy in both arms. | Duration of each cycle will be 28 or 21 days; patients will attend a follow-up visit 30 days after last study treatment. Follow-up for safety and efficacy will occur 6 months after the last patient is accrued to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Zhang, M.D., Study Director — Eisai Inc.
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - CTRC, San Antonio, Texas